CLINICAL TRIAL: NCT02805179
Title: Phase II Study of High Dose Radiotherapy and Concurrent Temozolomide Using Biologically-Based Target Volume Definition in Patients With Newly Diagnosed Glioblastoma
Brief Title: A Study of High-Dose Chemoradiation Using Biologically-Based Target Volume Definition in Patients With Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2012.006; HUM00113549 (Other: University of Michigan)
Record Dates: First submitted 2016-05-12; First posted 2016-06-17 (Estimated); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Dose Chemoradiation (Experimental): Patients will receive high dose radiation based in part on advanced imaging, and concurrent temozolomide. Four weeks after the completion of chemoradiation, patients will receive adjuvant temozolomide.
  Interventions: Radiation: High Dose Radiation; Drug: Temozolomide

INTERVENTIONS:
Radiation: High Dose Radiation — Radiation will be delivered once daily for a total of 30 fractions, five days per week.
Drug: Temozolomide — Patients will receive concurrent temozolomide (75 mg/m^2 daily for 6 weeks). Adjuvant temozolomide will be given at 150-200 mg/m^2, D1-5 every 28 days for a minimum of six cycles and will be started approximately four weeks following completion of radiotherapy.

SUMMARY:
This is a study to determine the safety and effectiveness of high-dose radiation therapy (RT) with concurrent temozolomide in patients with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
After analysis demonstrated the improved prognostic value of identifying both hypercellular tumor (TVHCV) based on high b-value diffusion-weighted magnetic resonance imaging (DW-MRI) and hyperperfused tumor (TVCBV) based on dynamic contrast-enhanced MRI (DCE-MRI), the study was amended and later-enrolled patients boosted to both TVHCV and TVCBV.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically-confirmed supratentorial World Health Organization (WHO) grade IV gliomas including glioblastoma multiforme and gliosarcoma
* Age 18 or older
* Karnofsky performance status (a measure to quantify general well being and activities of daily life; scale ranges from 0 to 100 where 100 is perfect health) of greater than or equal to 70
* Life expectancy of at least 12 weeks
* Adequate bone marrow reserve (hemoglobin greater than or equal to 10, absolute neutrophil count greater than or equal to 1500, platelets greater than or equal to 100,000); acceptable liver function (total bilirubin less than or equal to 2.0 mg/dl, ALT (Alanine Aminotransferase)/AST (Aspartate Aminotransferase) less than or equal to 5 times the normal range); acceptable renal function (serum creatinine less than or equal to 2.0 mg/dl). Eligibility level for hemoglobin may be reached by transfusion.
* Maximal contiguous volume of tumor based on high b-value diffusion MRI < 1/3 volume of brain
* Patients must be registered within 6 weeks of most recent resection.
* Patients must have signed a study-specific informed consent.

Exclusion Criteria:

* Recurrent glioma, or tumor involving the brainstem or cerebellum. Prior low-grade glioma without prior RT, now with malignant progression are eligible.
* Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment is not permitted. Prior chemotherapy for a different cancer is allowable, except for Temozolomide or Bevacizumab.
* Evidence of cerebrospinal fluid dissemination (positive cerebrospinal fluid cytology for malignancy or MRI findings consistent with CSF dissemination)
* Evidence of severe concurrent disease requiring treatment
* Prior invasive malignancy (except non-melanoma skin cancer) unless disease-free for a minimum of 3 years (for example, carcinoma in situ of breast, oral cavity or cervix are all permissible)
* Patients unable to undergo Magnetic Resonance Imaging exams (MRI) (i.e. patients with non-compatible devices such as cardiac pacemakers, other implanted electronic devices, metallic prostheses, or ferromagnetic prostheses (e.g. pins in artificial joints and surgical pins/clips) or unable to receive gadolinium for MRI, as per the standard UM Department of Radiology MRI screening criteria)
* Patients treated with previous cranial or head/neck radiotherapy leading to radiation field overlap
* Females of child-bearing potential must have a negative pregnancy test within 14 days prior to registration. Patients with reproductive potential must agree to use an effective contraceptive method during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kim, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Lee SW, Fraass BA, Marsh LH, Herbort K, Gebarski SS, Martel MK, Radany EH, Lichter AS, Sandler HM. Patterns of failure following high-dose 3-D conformal radiotherapy for high-grade astrocytomas: a quantitative dosimetric study. Int J Radiat Oncol Biol Phys. 1999 Jan 1;43(1):79-88. doi: 10.1016/s0360-3016(98)00266-1. PMID 9989517

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Patients will receive high dose radiation based in part on advanced imaging, and concurrent temozolomide. Four weeks after the completion of chemoradiation, patients will receive adjuvant temozolomide. High Dose Radiation: Radiation will be delivered once daily for a total of 30 fractions, five days per week. Temozolomide: Patients will receive concurrent temozolomide (75 mg/m^2 daily for 6 weeks). Adjuvant temozolomide will be given at 150-200 mg/m^2, D1-5 every 28 days for a minimum of six cycles and will be started approximately four weeks following completion of radiotherapy.
Period: Overall Study
Arm/Group | All Participants
Started | 26
Eligible Patients That Started Dose-intensified Chemo-radiation | 23
Subset of Participants, Boosted to Both High B-value Diffusion and Perfusion (Protocol amended to include perfusion) | 13
Completed | 23
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- High Dose Chemoradiation: Patients will receive high dose radiation based in part on advanced imaging, and concurrent temozolomide. Four weeks after the completion of chemoradiation, patients will receive adjuvant temozolomide. High Dose Radiation: Radiation will be delivered once daily for a total of 30 fractions, five days per week. Temozolomide: Patients will receive concurrent temozolomide (75 mg/m^2 daily for 6 weeks). Adjuvant temozolomide will be given at 150-200 mg/m^2, D1-5 every 28 days for a minimum of six cycles and will be started approximately four weeks following completion of radiotherapy.
Arm/Group | High Dose Chemoradiation
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: years] | 62 [50 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 12 Months
Description: Percentage of patients alive at 12 months after completion of chemoradiation
Time Frame: 12 months after completion of chemoradiation
Population: all eligible patients who completed dose-intensified chemo-radiation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Dose Chemoradiation
Number analyzed (Participants) | 23
percentage of participants
  all eligible patients who completed dose-intensified chemo-radiation | 74 [56 to 92]
  only patients who were boosted to both diffusion and perfusion: number analyzed (Participants) | 13
  only patients who were boosted to both diffusion and perfusion | 92 [78 to 100]
Statistical Analysis 1: Comparison: High Dose Chemoradiation; Test type: Superiority — Compared to historical controls; p = 0.03, 1-sided binomial test

2. Primary Outcome: Median Overall Survival
Description: Median overall survival in months
Time Frame: Median follow-up time was 26 months
Population: all eligible patients who completed dose-intensified chemo-radiation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | High Dose Chemoradiation
Number analyzed (Participants) | 23
months
  all eligible patients who completed dose-intensified chemo-radiation | 20 [14 to 29]
  only patients who were boosted to both diffusion and perfusion: number analyzed (Participants) | 13
  only patients who were boosted to both diffusion and perfusion | 20 [18 to NA] — Upper limit was not reached due to insufficient number of participants with events.

3. Secondary Outcome: Median Progression-free Survival
Description: From start of RT until disease progression or death, or until date of last imaging follow-up, estimated using Kaplan-Meier. Progression is defined by any of the following: >= 25% increase in sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids; a significant increase in T2/FLAIR non-enhancing lesions on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy, not due to comorbid events; appearance of any new lesions; clear progression of non-measurable lesions; or definite clinical deterioration not attributable to causes other than tumor, or to decrease in corticosteroid dose. When pathologic confirmation was unavailable, progression was defined as worsening enhancement based on imaging with or without adjunctive advanced imaging including perfusion MRI or magnetic resonance spectroscopy, when clinically indicated.
Time Frame: Median follow-up time was 26 months
Population: all eligible patients who completed dose-intensified chemo-radiation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | High Dose Chemoradiation
Number analyzed (Participants) | 23
months
  all eligible patients who completed dose-intensified chemo-radiation | 10 [7 to 17]
  only patients who were boosted to both diffusion and perfusion: number analyzed (Participants) | 13
  only patients who were boosted to both diffusion and perfusion | 12 [10 to 17]

4. Secondary Outcome: Median Change in Tumor Volume From Baseline to Mid-radiation Treatment (Week 4)
Description: Tumor volume will be measured by diffusion MRI and perfusion MRI before treatment start and at mid-treatment.
Time Frame: Baseline to Week 4
Population: All enrolled patients had available imaging were included in this analysis
Measure: Median (Inter-Quartile Range); unit: cubic centimeters
Arm/Group | High Dose Chemoradiation
Number analyzed (Participants) | 26
cubic centimeters | -2.9 [-5.3 to -1.8]

5. Secondary Outcome: Percentage of Patients That Experienced Deterioration in Quality of Life (QOL)
Description: Percentage of patients that experienced deterioration in QOL per the European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire (EORTC QLQ-C30). EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score=better level of physical functioning.
Time Frame: Baseline to 1 and 7 months
Population: all eligible patients who completed dose-intensified chemo-radiation
Measure: Number; unit: percentage of participants
Arm/Group | High Dose Chemoradiation
Number analyzed (Participants) | 23
percentage of participants
  at 1 month | 26
  at 7 months | 33

6. Secondary Outcome: Percentage of Patients With Failure; Central or In-field vs. Marginal or Distant
Description: Failures will be classified as central or in-field, marginal or distant based on previously published criteria. 1) "central," in which 95% or more of the recurrent tumor volume (Vrecur) was within D95, the region treated to high dose (95% of the prescription dose); 2) "in-field," in which 80% or more of Vrecur was within the D95 isodose surface; 3) "marginal," when between 20 and 80% of Vrecur was inside the D95 surface; 4) "outside," in which less than 20% of Vrecur was inside the D95 surface.
Time Frame: Median 26 months
Population: all eligible patients who completed dose-intensified chemo-radiation
Measure: Number; unit: percentage of participants
Arm/Group | High Dose Chemoradiation
Number analyzed (Participants) | 23
percentage of participants
  central or in-field | 31
  non-central/non-in-field (marginal or distant) | 69

ADVERSE EVENTS:
Time Frame: Time frame for toxicity was from the time of the initial intervention through 30 days following the completion of radiation therapy. Subacute and late neurologic toxicity beyond 30 days was assessed every 2 to 3 months, and all patients were monitored for late neurologic toxicity until last follow-up or death. The median follow-up time was 26 months.
Groups:
- All Enrolled Patients: Patients will receive high dose radiation based in part on advanced imaging, and concurrent temozolomide. Four weeks after the completion of chemoradiation, patients will receive adjuvant temozolomide. High Dose Radiation: Radiation will be delivered once daily for a total of 30 fractions, five days per week. Temozolomide: Patients will receive concurrent temozolomide (75 mg/m^2 daily for 6 weeks). Adjuvant temozolomide will be given at 150-200 mg/m^2, D1-5 every 28 days for a minimum of six cycles and will be started approximately four weeks following completion of radiotherapy.
Arm/Group | All Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 21/26
Serious Adverse Events (participants affected / at risk) | 8/26
Other Adverse Events (participants affected / at risk) | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Patients (N=26)
Nausea (Gastrointestinal disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 2 (3)
Confusion (Psychiatric disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Patients (N=26)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Eye disorders - Other (Eye disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (15)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 20 (26)
Gait disturbance (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 5 (7)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 5 (6)
Allergic reaction (Immune system disorders) | 3 (4)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Investigations - Other (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 7 (16)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7)
Dysarthria (Nervous system disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 8 (8)
Hypersomnia (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 4 (6)
Seizure (Nervous system disorders) | 3 (4)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 7 (9)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT02805179/Prot_SAP_000.pdf